CLINICAL TRIAL: NCT00534820
Title: Cytogenetic Analysis of Bone Marrow Specimen Prior to High Dose Chemotherapy and Autologous Stem Cell Transplantation in Patients With Non-Hodgkin's Lymphoma or Hodgkin's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RAC#2041015
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Cytogenetic Analysis of Bone Marrow Specimen in Non-Hodgkin's Lymphoma or Hodgkin's Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cytogenetic Analysis of Bone Marrow Specimen — Cytogenetic Analysis of BM Specimen

SUMMARY:
Cytogenetic Analysis of Bone Marrow Specimen Prior to High Dose Chemotherapy and Autologous Stem Cell Transplantation in Patients with Non-Hodgkin's Lymphoma or Hodgkin's Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non-Hodgkin's Lymphoma or Hodgkin's Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2004-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Syed Akhtar, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia